CLINICAL TRIAL: NCT06203028
Title: Investigation of the Effectiveness of Cyberbullying Awareness Training Given to Secondary School Students
Brief Title: Cyberbullying Awareness Training for Secondary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Emine Ekici, Assistant Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/17-14
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Cyberbullying
Keywords: cyberbullying; students; school
MeSH Terms: conditions — Cyberbullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The 'Cyberbullying Awareness Training' program will be implemented in 2 sessions in 1 day for a total of 2 hours.
  Interventions: Behavioral: Cyberbullying Awareness Training
- Control Group (No Intervention): The Cyberbullying Awareness Training program will not be applied to students in the control group.

INTERVENTIONS:
Behavioral: Cyberbullying Awareness Training — The 'Cyberbullying Awareness Training' program will be implemented in 2 sessions in 1 day for a total of 2 hours. The training program will be implemented in line with the headings 'Definition of cyberbullying, Cyberbullying tools and practices, Case studies on cyberbullying, Causes of cyberbullying, Academic, social, psychological and physical effects of cyberbullying, Coping strategies with cyberbullying'.
  Arms: Experimental Group

SUMMARY:
The study will be conducted with the randomized controlled experimental method. The purpose of this research is to determine the cyberbullying awareness training given to 7th-grade secondary school students' awareness levels of cyberbullying. Students will be randomly assigned to groups by lottery method. After the randomization students in the intervention group will be given 'Cyberbullying Awareness Training'. The cyberbullying awareness level of all students will be determined with the 'Cyberbullying Awareness Scale' before and 3 months after the training. Students in the control group will not be educated. The cyberbullying awareness level of the students in the control group will be determined with the 'Cyberbullying Awareness Scale' when they are included in the research and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 12 and 14,
* No auditory, visual, or mental problems that would affect communication
* Speaking and understanding Turkish at native level

Exclusion Criteria:

* Being younger than 12 years old and older than 14 years old,
* Having auditory, visual, or mental problems that would affect communication
* Not speaking and understanding Turkish at native level

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Cyberbullying Awareness Level | Before and 3 months after the Cyberbullying Awareness Training.
  "Cyberbullying Awareness Scale" will be used to determine students' cyberbullying awareness levels. Regarding the consistency of the scale, Cronbach's alpha value was found to be 0.89. As a result of the clustering analysis, it was found appropriate to cluster the total score to be obtained from the scale as 21-61, 62-81, 82-105, and it was stated that the score range of 21-61 can be expressed as low, 62-81 as medium and 82-105 as high cyberbullying awareness. Those who will fill in the cyberbullying awareness scale mark their level of agreement with each statement in the scale between the options (1) strongly disagree and (5) strongly agree. A minimum score of 21 and a maximum score of 105 can be obtained from the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Erkut, PhD, Principal Investigator — Maltepe Üniversitesi Hemşirelik Yüksekokulu
Locations (1):
- Maltepe University, Istanbul, İ̇stanbul, Turkey (Türkiye)